CLINICAL TRIAL: NCT00671853
Title: Quetiapine XR in the Treatment of Comorbid Generalized Anxiety Disorder in Bipolar Depression With or Without Substance Use Disorder
Brief Title: Quetiapine Extended Release (XR) in Bipolar Patients With Comorbid Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood & Anxiety Clinic, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-06-19
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Disorder; Anxiety; Anxiety Disorders; Substance Use Disorders
Keywords: Bipolar Disorder; Anxiety; Anxiety Disorders; Substance Use Disorders
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine XR
  Interventions: Drug: Quetiapine XR
- 2 (Placebo Comparator): Placebo for quetiapine XR
  Interventions: Drug: Placebo for quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — Days 1-2 - 50 mg/day; Days 3-4 - 150mg/day; Day 5-End of Study - 300mg/day
  Other Names: Seroquel XR
  Arms: 1
Drug: Placebo for quetiapine XR — Days 1-2 - 50 mg/day; Days 3-4 - 150mg/day; Day 5-End of Study - 300mg/day
  Other Names: Placebo for Seroquel XR
  Arms: 2

SUMMARY:
The primary objective is to test the hypothesis that Quetiapine XR (Extended Release) monotherapy and adjunctive therapy is effective in the acute treatment of bipolar depression and comorbid generalized anxiety disorder in patients with bipolar disorder with or without a substance use disorder. The secondary aim is to generate an estimate of effect size to power a definitive large-scale, multi-site collaborative R01 and to configure the use of the primary and secondary outcome measures in the definitive large-scale study.

DETAILED DESCRIPTION:
120 subjects aged 18 and up with Diagnostic and Statistical Manual -IV Generalized Anxiety Disorder and Bipolar Disorder type I or II as identified by extensive clinical interview and the Mini-International Neuropsychiatric Interview (MINI) will be enrolled and randomized. Assignment to each arm will be balanced for BP I vs BP II; male vs female; and with vs without SUD. Potential participants will be recruited by means of Institutional Review Board -approved advertising or from the clinical psychiatric infrastructure.

This study is a randomized, double-blind, placebo-controlled, 8-week comparison of quetiapine sustained-release monotherapy or adjunctive mood stabilizer therapy vs. placebo in the acute treatment of comorbid generalized anxiety disorder in patients with bipolar disorder with or without a substance use disorder. Subjects will be assessed weekly for mood changes and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV diagnosis of bipolar I or II disorder, and currently depressed as confirmed by the MINI-Plus at Screening.
* Diagnostic and Statistical Manual-IV diagnosis of lifetime GAD;
* Hamilton Depression Rating Scale -17 items total score ≥ 18;
* Hamilton Anxiety Rating Scale total score ≥ 18;
* Be male or female at least 18 year old and not older than 65.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Severe medical or neurological problems.
* Severe personality disorder.
* Currently suicidal risk judged by physician.
* Known history of intolerance or hypersensitivity to any of the medications involved in the study.
* Treatment with quetiapine at any dose in the 6 months prior to randomization.
* Known lack of response to quetiapine in a dosage of at least 50 mg for 4 weeks at any time, as judged by the investigator.
* Dependence on opiate, phencyclidine (PCP), and/or barbiturate.
* Acute mania as determined by a score > 12 on the Young Mania Rating Scale at baseline.
* Concurrent obsessive compulsive disorder.
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrolment or randomisation of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
* A patient with diabetes mellitus (DM) fulfilling one of the following criteria: a. Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) .8.5% b. Admitted to hospital for treatment of DM or DM related illness within the past 12 weeks c. Not under physician care for DM d. Physician responsible for patient's DM care has not indicated that the patient's DM is controlled f. Physician responsible for patient's DM care has not approved the patient's participation in the study g. Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks before randomization. For thiazolidinediones (glitazones) this period should not be less than 8 weeks before randomization h. Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a patient with DM meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, PhD, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gao K, Wu R, Kemp DE, Chen J, Karberg E, Conroy C, Chan P, Ren M, Serrano MB, Ganocy SJ, Calabrese JR. Efficacy and safety of quetiapine-XR as monotherapy or adjunctive therapy to a mood stabilizer in acute bipolar depression with generalized anxiety disorder and other comorbidities: a randomized, placebo-controlled trial. J Clin Psychiatry. 2014 Oct;75(10):1062-8. doi: 10.4088/JCP.13m08847. PMID 25007003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consent 120 subjects. However, 29 subjects were considered screening failures and were not randomized.
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Started | 46 | 45
Completed | 26 | 18
Not Completed | 20 | 27
Not completed — Lack of Efficacy | 3 | 7
Not completed — Adverse Event | 7 | 1
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 8 | 8
Not completed — Physician Decision | 0 | 2
Not completed — Non-adherence with study procedures | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 45 | 91
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (12) | 37.4 (11.3) | 37.7 (11.6)
Gender [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change in the 17 Item Hamilton Rating Scale for Depression (HAM-D-17) Score
Description: A score of 0-7 is considered to be normal. Hamilton Rating Scale total score ranges from 0-57 where higher scores are indicative of more depression.
Time Frame: Week 0 - Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
units on a scale | -9.91 (16.45) | -7.41 (8.13)

2. Secondary Outcome: Response Rate (≥ 50% Improvement) on Hamilton Rating Scale for Depression (HAM-D-17)
Description: as for outcome 1
Time Frame: Week 0 - Week 8
Measure: Number; unit: participants
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
participants | 12 | 11

3. Secondary Outcome: Remission Rate (≤ 7) on Hamilton Rating Scale for Depression (HAM-D-17)
Description: A score of 0-7 is considered to be normal. Hamilton Rating Scale total score ranges from 0-57 where higher scores are indicative of more depression. Remission is defined by the number of participants with Hamilton Rating Scale for Depression score equal to or less than 7.
Time Frame: Week 0 - Week 8
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
Participants | 6 | 6

4. Secondary Outcome: Change in Clinical Global Impressions of Improvement or Severity (CGI-I or S) Score
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment.
  1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Week 0 - Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
units on a scale | -1.10 (1.16) | -0.8 (1.21)

5. Secondary Outcome: Change in the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Score
Description: This assessment degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70 with a higher score indicating less enjoyment and satisfaction.
Time Frame: Week 0 - Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
units on a scale | 0.11 (0.22) | -0.06 (0.52)

6. Secondary Outcome: Change in Hamilton Rating Scale for Anxiety (HAM-A)
Description: The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe
Time Frame: Week 0 - Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Number analyzed (Participants) | 46 | 45
units on a scale | -9.54 (7.58) | -8.25 (8.70)

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo for Quetiapine XR
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 44/46 | 37/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine XR (N=46) | Placebo for Quetiapine XR (N=45)
Dry Mouth (Ear and labyrinth disorders) | 27 (27) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Stomach Upset (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dizziness (General disorders) | 8 (8) | 8 (8)
Headache (General disorders) | 7 (7) | 3 (3)
Increased Appetite (General disorders) | 1 (1) | 4 (4)
Sedation (Psychiatric disorders) | 4 (4) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes